CLINICAL TRIAL: NCT01956838
Title: The Effect of Bitter, Umami and Sweet Tastants on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL44428.068.13/METC 13-2-025
Record Dates: First submitted 2013-09-17; First posted 2013-10-08 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
Keywords: food intake; tastants; obesity
MeSH Terms: conditions — Obesity | interventions — Candy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Umami (Experimental): intraduodenal infusion of umami
  Interventions: Dietary Supplement: umami
- sweet (Experimental): intraduodenal infusion of sweet tastant
  Interventions: Dietary Supplement: sweet
- bitter (Experimental): intraduodenal infusion of bitter tastant
  Interventions: Dietary Supplement: bitter
- combination (Experimental): intraduodenal infusion of a combination of tastants (umami, bitter and sweet)
  Interventions: Dietary Supplement: umami; Dietary Supplement: bitter; Dietary Supplement: sweet
- placebo (Placebo Comparator): intraduodenal infusion of placebo (tap water)

INTERVENTIONS:
Dietary Supplement: umami — intraduodenal infusion of umami tastant
  Arms: Umami; combination
Dietary Supplement: bitter — intraduodenal infusion of bitter tastant
  Arms: bitter; combination
Dietary Supplement: sweet — intraduodenal infusion of sweet tastant
  Arms: combination; sweet

SUMMARY:
Rationale: The appearance of tastants in the small intestine can result in the activation of a negative feedback mechanism from different parts of the intestine to the stomach, the small intestine and to the central nervous system. These processes inhibit food processing, appetite sensations and food intake, and furthermore they increase feelings of satiety and satiation. We will investigate the effects of intraduodenal infusion of quinine 75mg (bitter), rebaudioside A 540mg (sweet), monosodium glutamate 2g (umami), a combination of these tastants (quinine, rebaudioside A, monosodium glutamate) and placebo (5 test days in total) on ad libitum food intake, satiation and in vivo release of the gut satiety peptides CCK and GLP-1.

Study design: To assess the effect of intraduodenal infusion of single ingredients and a combination of tastants (bitter, umami and sweet) on ad libitum food intake.

Secondary Objective(s):

1. To investigate the effect of intraduodenal delivery of a combination of tastants on satiation.
2. To assess the effect of intraduodenal delivery of a combination of tastants on gastrointestinal hormone release.
3. To assess the effects of the tastants quinine, rebaudioside A and monosodium glutamate on the parameters as mentioned under the primary objective, and under secondary objectives 1 and 2.
4. To compare the effects, as mentioned under the primary objective, and under secondary objectives 1 and 2, of the combination of tastants to those of the three single tastants quinine, rebaudioside A and monosodium glutamate.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years. This study will include healthy adult subjects (male and female). Women must be taking contraceptives.
* BMI between 18 and 25 kg/m2)
* Weight stable over at least the last 6 months

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Blood donation within 3 months before the study period
* Self-admitted HIV-positive state
* Weight <60kg
* Non-tasters of sweet, bitter or umami
* Evidence of MSG-hypersensitivity or Chinese restaurant syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Ad libitum meal intake | 5 weeks
  Difference in ad libitum meal intake (as measured during ad libitum pasta meal). At end of the testday

SECONDARY OUTCOMES:
Satiation | 5 weeks
  Difference in satiation (as measured by VAS) per time point
Gut hormones | 5 weeks
  Measurements in plasma levels of the gut hormones CCK, GLP-1, insulin and glucose

CONTACTS AND LOCATIONS:
Overall Officials: Prof Masclee, MD,PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] van Avesaat M, Troost FJ, Ripken D, Peters J, Hendriks HF, Masclee AA. Intraduodenal infusion of a combination of tastants decreases food intake in humans. Am J Clin Nutr. 2015 Oct;102(4):729-35. doi: 10.3945/ajcn.115.113266. Epub 2015 Aug 19. PMID 26289437